CLINICAL TRIAL: NCT01200485
Title: A Randomized Phase 2 Study to Evaluate the Efficacy of Rasburicase in Patients at Risk for TLS During Two Cycles of Chemotherapy
Brief Title: Rasburicase in Patients at High Risk for Tumor Lysis Syndrome (TLS) During Cycle-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0284; NCI-2012-01889 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Results first posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Leukemia; Lymphoma
Keywords: Supportive Care; Recombinant urate oxidase; Chemotherapy; Tumor Lysis Syndrome (TLS); Hematologic malignancies; Acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Lymphoma; Tumor Lysis Syndrome; Hematologic Neoplasms; Leukemia, Myeloid, Acute | interventions — rasburicase; Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Rasburicase Alone (Experimental): Rasburicase by vein on Day 1 (0.15 mg/kg or a flat dose of 3 mg) as a single dose, plus as needed dosing (until day 5), during cycle 1 (21 day cycle).
  Interventions: Drug: Rasburicase
- Arm A (Rasburicase) (Experimental): Participants randomized to Rasburicase (0.15 mg/kg) by vein on day 1 plus as needed dosing (until day 5) during Cycle 2.
  Interventions: Drug: Rasburicase
- Arm B (Allopurinol) (Experimental): Participants randomized to Allopurinol (300 mg/day) by vein each day on Days 1-5 of Cycle 2.
  Interventions: Drug: Allopurinol

INTERVENTIONS:
Drug: Rasburicase — Cycle 1: 3 mg/kg by vein on Day 1, plus as needed dosing (until day 5), during Cycle 1.
  Cycle 2 Arm A: 0.15 mg/kg by vein on Day 1 of Cycle 2, plus as needed dosing (until day 5), during Cycle 2.
  Arms: Arm A (Rasburicase); Rasburicase Alone
Drug: Allopurinol — Arm B: 300 mg/day by vein, as standard of care, over 30 minutes each day on days 1-5 of cycle 2 in 21 day cycle.
  Other Names: Loprin; Zurinol; Zyloprim
  Arms: Arm B (Allopurinol)

SUMMARY:
The goal of this clinical research study is to learn if using Elitek (rasburicase) for 2 cycles can help to control or prevent TLS better than 1 cycle of rasburicase and 1 cycle of allopurinol. The safety of this treatment will also be studied.

DETAILED DESCRIPTION:
Study Drugs:

Rasburicase is designed to help decrease or prevent the high level of uric acid that may occur during the beginning of chemotherapy. A high level of uric acid results from TLS and can lead to kidney failure.

Allopurinol is designed to help block uric acid. It is the standard of care for helping to control increased uric acid levels caused by TLS.

Study Groups and Drug Administration:

Each cycle will last about 3 weeks.

If you are found to be eligible to take part in this study, you will receive rasburicase by vein over about 30 minutes on Day 1 of Cycle 1 (about 4 hours before you begin receiving chemotherapy). If the doctor thinks it is needed, you may also receive the drug on Days 2-5 of Cycle 1.

For Cycle 2, you will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups. There is an equal chance of being assigned to either group:

* If you are in Group A, you will receive rasburicase on Day 1 of Cycle 2. If the doctor thinks it is needed, you may also receive the drug on Days 2-5 of Cycle 2.
* If you are in Group B, you will receive allopurinol by vein over 30 minutes each day on Days 1-5 of Cycle 2.

Group B Participants: If your uric acid blood levels continue to increase in Cycle 2 and you show symptoms of tumor lysis syndrome, you may receive rasburicase as a single dose. If the doctor thinks it is needed, you may also receive 1 or more additional dose(s).

Study Visits:

On Day 1 of Cycle 1:

* Blood (about 1 teaspoon) will be drawn to check uric acid levels before and 4 hours after you receive rasburicase.
* Blood (about 2 tablespoons) will be drawn for routine tests.
* Blood (about 1 teaspoon) will be drawn for antibody testing. Antibodies are proteins made by the body that the immune system uses to help prevent disease.

On Days 2-5 of Cycle 1:

* Blood (about 1 teaspoon) will be drawn to check uric acid levels.
* Blood (about 2 tablespoon) will be drawn for routine tests.

At the end of both cycles, blood (about 1 teaspoon) will be drawn for antibody testing.

Length of Study:

You will receive drugs on this study for up to 2 cycles. You will be taken off study if intolerable side effects occur.

Your participation in the study will be over after the follow-up visit.

Follow-Up:

Three (3) months after the end of Cycle 2, blood (about 1 teaspoon) will be drawn for antibody testing.

This is an investigational study. Allopurinol is commercially available and FDA approved to treat TLS. Rasburicase is commercially available and FDA approved for treating TLS for 1 cycle in patients with leukemia, lymphoma, and solid tumor cancers who are receiving anti-cancer therapy. It is investigational to give rasburicase for 2 cycles.

Up to 55 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients that are high risk for TLS or potential/intermediate risk for TLS as described below: (a) High risk: Hyperuricemia of malignancy (Uric acid levels >7.5); or diagnosis of very aggressive lymphoma/leukemia based on Revised European-American Lymphoma (REAL) classification; acute myeloid leukemia, CML in blast crisis; high grade myelodysplastic syndrome only if they have >10% bone marrow blast involvement and given aggressive treatment similar to acute myeloid leukemia (AML). (b) Potential risk: Diagnosis of aggressive lymphoma/leukemia based on (REAL) classification. Plus one or more of the following criteria: lactate dehydrogenase (LDH) >/= 2 x upper limit of normal (UNL); Stage III-IV disease; Stage I-II disease with at least 1 lymph node/tumor > 5 cm in diameter. For patients with potential/intermediate risk for TLS- Only those planned to receive alternating regimens (or non-standard regimens) in 2 cycles (example; R-Hyper-central venous access device (CVAD) alternating with MTX/ARA-C) will be eligible.
2. Eastern Cooperative Oncology Group (ECOG) performance status 0-3.
3. Negative pregnancy test (females of child bearing potential) within </= 1 week of rasburicase dose and use of efficient contraceptive method (both males and females). Pregnancy test may be performed on serum (HCG) or urine (HCG).
4. Signed written informed consent approved by the Institutional Review Board obtained prior to study entry.

Exclusion Criteria:

1. Prior H/O severe allergy or asthma requiring active treatment.
2. Patients with mantle cell lymphoma (MCL) with stage 1 or 2 disease.
3. Patient receiving any investigational drug for hyperuricemia within 30 days of planned first treatment with rasburicase.
4. Pregnancy or lactation.
5. Known history of glucose-6-phosphate dehydrogenase (G6PD) deficiency.
6. Known history of hemolysis and/or methemoglobinemia.
7. Previous therapy with urate oxidase.
8. Conditions unsuitable for participation in the trial in the Investigator's opinion.
9. Unwillingness to comply with the requirements of the protocol.
10. Use of allopurinol within 72 hours of the study entry.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2011-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saroj Vadhan-Raj, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: April 25, 2011 to September 10, 2015. All recruitment done at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: Cycle 2 is the study cycle; of the 55 participants enrolled on study, 52 were treated in cycle 1 (rasburicase alone), and only 46 were randomized onto the two arms in the study cycle (cycle 2, Arm A: Rasburicase; Arm B: Allopurinol).
Groups:
- Cycle 1: Rasburicase Alone: Rasburicase by vein on Day 1 (0.15 mg/kg or a flat dose of 3 mg) as a single dose, plus as needed dosing (until day 5), during cycle 1 (21 day cycle).
- Cycle 2, Arm A: Rasburicase: Rasburicase (0.15 mg/kg) by vein on day 1 plus as needed dosing (until day 5) during Cycle 2.
- Cycle 2, Arm B: Allopurinol: Allopurinol (300 mg/day) each day on Days 1-5 of Cycle 2.
Period: Cycle 1: Rasburicase Alone Delivery
Arm/Group | Cycle 1: Rasburicase Alone | Cycle 2, Arm A: Rasburicase | Cycle 2, Arm B: Allopurinol
Started | 55 (Of 55 participants screened, only 52 treated.) | 0 | 0
Completed | 52 | 0 | 0
Not Completed | 3 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Insurance Coverage Denied | 2 | 0 | 0
Period: Cycle 2: Randomization
Arm/Group | Cycle 1: Rasburicase Alone | Cycle 2, Arm A: Rasburicase | Cycle 2, Arm B: Allopurinol
Started | 0 (Of 55 enrolled on study, 52 participants were treated in Cycle 1, only 46 randomized to Cycle 2) | 21 (Six not randomized: Methemoglobinemia-1, Kidney failure-2, Chemotherapy changed-2, Not evaluable-1) | 25
Completed | 0 | 21 | 25
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Of 55 enrolled on study, 52 participants were treated in Cycle 1 Rasburicase alone, only 46 randomized to Cycle 2 Arm A Rasburicase (21) and Arm B Allopurinol (25).
Groups:
- Rasburicase Alone: Rasburicase by vein on Day 1 (0.15 mg/kg or a flat dose of 3 mg) as a single dose, plus as needed dosing (until day 5), during cycle 1
Arm/Group | Rasburicase Alone
Number analyzed (Participants) | 55
Age, Continuous [Median (Full Range); unit: years] | 54 [24 to 78]
Age, Customized [Median (Full Range); unit: years] — Baseline age of participants randomized in Cycle 2. Population: Each row represents continuous age for each randomized arm in Cycle 2, Arm A Rasburicase (N=21) and Arm B Allopurinol (N=25), total 46.
  years
    Cycle 2, Arm A: number analyzed (Participants) | 21
    Cycle 2, Arm A | 52 [30 to 75]
    Cycle 2, Arm B: number analyzed (Participants) | 25
    Cycle 2, Arm B | 56 [24 to 76]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Measure rows divide Cycle 1 (55) then those randomized to Cycle 2 Arm A (21) and Arm B (25).
  Participants
    Cycle 1, Rasburicase: Female | 15
    Cycle 1, Rasburicase: Male | 40
    Cycle 2, Arm A: number analyzed (Participants) | 21
    Cycle 2, Arm A: Female | 5
    Cycle 2, Arm A: Male | 16
    Cycle 2, Arm B: number analyzed (Participants) | 25
    Cycle 2, Arm B: Female | 8
    Cycle 2, Arm B: Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 55
Eastern Cooperative Oncology Group (ECOG) PS, Cycle 1 [Number; unit: participants] — Participant performance status (PS) using the ECOG scale which ranges from 0 to 4, with 0 being fully functional and asymptomatic, and 4 being bedridden.
  participants
    <2 | 53
    >/=2 | 2
ECOG PS, Cycle 2 [Count of Participants; unit: Participants] — Row represents PS as defined above for each randomized arm in Cycle 2, Arm A (21) and Arm B (25), total 46. Population: Randomized arms in Cycle 2 Arm A (21) and Arm B (25).
  Participants
    Arm A: number analyzed (Participants) | 21
    Arm A: <2 | 20
    Arm A: >/=2 | 1
    Arm B: number analyzed (Participants) | 25
    Arm B: <2 | 24
    Arm B: >/=2 | 1
Tumor Lysis Syndrome (TLS) Risk [Count of Participants; unit: Participants] — High risk: Hyperuricemia of malignancy (Uric acid level>7.5); or diagnosis aggressive lymphoma/leukemia based on Revised European-American Lymphoma (REAL) classification; acute myeloid leukemia, CML in blast crisis; high grade myelodysplastic syndrome only if >10% bone marrow blast involvement, aggressive treatment similar to acute myeloid leukemia (AML). Potential risk: Diagnosis aggressive lymphoma/leukemia (REAL classification) + 1/> criteria: lactate dehydrogenase (LDH) >2 x upper limit of normal (UNL); Stage III-IV disease; Stage I-II disease + 1/> lymph node/tumor >5 cm diameter.
  Participants
    High | 22
    Potential | 30
    Not evaluable | 3
Baseline Plasma Uric Acid (PUA) [Count of Participants; unit: Participants] — PUA determined by uric acid blood test. Population: Randomized Cycle 2 Arm A (21) and Arm B (25).
  Participants
    Arm A: number analyzed (Participants) | 21
    Arm A: <7.1 mg/dL | 16
    Arm A: >/=7.1 mg/dL | 4
    Arm A: Not evaluated | 1
    Arm B: number analyzed (Participants) | 25
    Arm B: <7.1 mg/dL | 22
    Arm B: >/=7.1 mg/dL | 3
    Arm B: Not evaluated | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants (Incidence) of LTLS (Laboratory Tumor Lysis Syndrome)
Description: Number of participants (incidence) of LTLS in the two arms, as defined by the Cairo-Bishop criteria , during cycle 2.
  Cairo-Bishop criteria:
  Uric acid x ≥ 476 μmol/l or 25% increase from baseline Potassium x ≥ 6·0 mmol/l or 25% increase from baseline Phosphorous x ≥ 2·1 mmol/l (children), x ≥1·45 mmol/l (adults) or 25% increase from baseline Calcium x ≤ 1·75 mmol/l or 25% decrease from baseline Laboratory tumour lysis syndrome (LTLS) is defined as either a 25% change or level above or below normal, as defined above, for any two or more serum values of uric acid, potassium, phosphate, and calcium within 3d before or 7d after the initiation of chemotherapy.
Time Frame: Up to two 3-week cycles, 6 weeks
Population: All 46 participants treated in randomized cycle 2 of study were included in analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Arm A (Rasburicase): Rasburicase (0.15 mg/kg) by vein on day 1 plus as needed dosing (until day 5) during Cycle 2.
- Arm B (Allopurinol): Allopurinol (300 mg/day) each day on Days 1-5 of Cycle 2.
Arm/Group | Arm A (Rasburicase) | Arm B (Allopurinol)
Number analyzed (Participants) | 21 | 25
Participants | 1 | 1

2. Primary Outcome: Number of Cycle 2 Participants Normalizing Uric Acid Levels (UAL) Within 24 Hours of Treatment
Description: Number of participants with normalized UAL as determined by a uric acid blood test at either 24 hours. A uric acid blood test, also known as a serum uric acid measurement, determines how much uric acid is present in the blood where normal levels are 2.4-6.0 mg/dL (female) and 3.4-7.0 mg/dL (male).
Time Frame: Up to 24 hours of cycle 2 dose delivery
Population: One participant in Arm A missed one UA level assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Rasburicase) | Arm B (Allopurinol)
Number analyzed (Participants) | 21 | 25
Participants | 20 | 25

ADVERSE EVENTS:
Time Frame: Adverse events were captured before and after each cycle, up to 30 days from day 1 of the study drug and clinical assessment
Groups:
- Cycle 2: Arm A (Rasburicase): Rasburicase (0.15 mg/kg) by vein on day 1 plus as needed dosing (until day 5) during Cycle 2.
- Cycle 2: Arm B (Allopurinol): Allopurinol (300 mg/day) each day on Days 1-5 of Cycle 2.
Arm/Group | Cycle 1: Rasburicase Alone | Cycle 2: Arm A (Rasburicase) | Cycle 2: Arm B (Allopurinol)
All-Cause Mortality (participants affected / at risk) | 0/52 | 1/21 | 1/25
Serious Adverse Events (participants affected / at risk) | 3/52 | 1/21 | 1/25
Other Adverse Events (participants affected / at risk) | 38/52 | 12/21 | 17/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cycle 1: Rasburicase Alone (N=52) | Cycle 2: Arm A (Rasburicase) (N=21) | Cycle 2: Arm B (Allopurinol) (N=25)
Death (General disorders) | 0 (0) | 1 (1) | 1 (1)
Methemoglobinemia (Blood and lymphatic system disorders) | 1 (1) | 0 | 0
Acute renal failure (Renal and urinary disorders) | 2 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cycle 1: Rasburicase Alone (N=52) | Cycle 2: Arm A (Rasburicase) (N=21) | Cycle 2: Arm B (Allopurinol) (N=25)
Fatigue (General disorders) | 21 | 9 (9) | 8 (8)
Headache (Nervous system disorders) | 10 | 4 (4) | 10 (10)
Constipation (Gastrointestinal disorders) | 23 | 4 (4) | 9 (9)
Blood bilirubin increased (Investigations) | 6 | 1 (1) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes